CLINICAL TRIAL: NCT02446353
Title: A Randomized, Open Label, Single Dose, Cross-over, Phase I Trial to Investigate Safety and Pharmacokinetics of Apetrol ES and Megace® Under Fasting and Fed Conditions in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Safety Study of Apetrol ES
Acronym: Apetrol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-ESCL001
Record Dates: First submitted 2015-05-07; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Male Volunteers
MeSH Terms: interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Megace : fed (Experimental): Megace / Apetrol ES : comparator / test, fed
  Interventions: Drug: Apetrol ES / Megace
- Apetrol ES : fed (Experimental): Apetrol ES / Megace : test / comparator, fed, cross-over
  Interventions: Drug: Apetrol ES / Megace
- Megace : fasting (Experimental): Megace / Apetrol ES : comparator / test, fasting
  Interventions: Drug: Apetrol ES / Megace
- Apetrol ES : fasting (Experimental): Apetrol ES / Megace : test / comparator, fasting, cross-over
  Interventions: Drug: Apetrol ES / Megace

INTERVENTIONS:
Drug: Apetrol ES / Megace — Sequences of administered drugs
  Other Names: Apetrol ES(ES81) 625 mg / 5mL, Megace 800mg / 20mL

SUMMARY:
A Randomized, Open Label, Single dose, Cross-over, Phase I Trial to Investigate Safety and Pharmacokinetics of Apetrol ES and Megace® in Healthy Male Volunteers.

DETAILED DESCRIPTION:
[Part 1] fasting [Part 2] fed

ELIGIBILITY:
Inclusion Criteria:

* Is a healty male between 20 and 55 years old.
* In a ± 20% than ideal body weight. [ideal body weight(kg) = height(cm)-100) x 0.9 (Broca's rule)
* Subjects who are considered to be suitable in conducting the clinical trial in serum test, hematology test, hemato-chemical test, urine test and 12-ECG result.
* Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Agrees to use an adequate means of contraception during clinical trials
* Subject who has voluntarily decided to participate in this clinical trial and consented in writing.

Exclusion Criteria:

* Is allergic against Megestrol acetate or other drugs (Aspirin, NSAIDs, Antibiotics, etc.) or against foods, or has an clinically serious allergic history.
* Subjects who have present condition or past history of any disease involving liver, kidney, nervous system, immune system, respiratory system, or endocrine system; hematologic and oncologic disease; cardiovascular disease; or psychiatric disorder (mood disorder, obsessive-compulsive disorder, etc. that may affect ADME of investigational medicinal products.
* In the vital signs measured in sitting position at the screening visit, subjects who have hypertension desease(a systolic blood pressure of ≥ 150 mmHg or a diastolic blood pressure of ≥ 100 mmHg).
* Diabetic patients or the patients who are abnormal of impaired glucose tolerance.
* The patients who have a history of Arterial Embolism.
* The patients who have a history of adrenal insufficiency like hypotension or nausea or vertigo or asthenia or etc.
* Subjects who have a history of drug abuse or shown positive reaction to drugs that may be abused from a urine drug screening
* Subjects who took any specialized drug or an herbal medication within 2 weeks before the date of first administration or took any over the counter (OTC) drug within 1 week (however, they may be included as subjects if appropriate depending on the investigator's discretion)
* Subjects who had whole blood donation within 2 months or component blood donation within 1 month before the clinical trial.
* Subjects who have abnormal diets that may affect ADME of investigational medicinal products.
* Subjects who have been drinking extremely alcohol and caffeine (more than caffeine 5 cups/day, soju 3 cups/day, beer 3 cups/day, liquors 2 cups/day, 10 cigarettes/day) or can't refrain from drinking during the clinical trial period.
* Subjects who had administration a barbiturates within 1 month before the date of first drug administration
* Subjects who already participated in other clinical trials within 2 months before this clinical trial.
* Subjects who are considered to be unsuitable in conducting the clinical trial for other reason at the principal investigator's discretionary judgment

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose(0h), 1, 2, 3, 4, 5, 6, (7), 8, 10, 12, 24, 48, 72, 96, 120 h
  16 times(fasting), 15 times(fed)
AUClast | Pre-dose(0h), 1, 2, 3, 4, 5, 6, (7), 8, 10, 12, 24, 48, 72, 96, 120 h
  16 times(fasting), 15 times(fed)

SECONDARY OUTCOMES:
AUCinf, %AUCextra | Pre-dose(0h), 1, 2, 3, 4, 5, 6, (7), 8, 10, 12, 24, 48, 72, 96, 120 h
  16 times(fasting), 15 times(fed)
Tmax | Pre-dose(0h), 1, 2, 3, 4, 5, 6, (7), 8, 10, 12, 24, 48, 72, 96, 120 h
  16 times(fasting), 15 times(fed)
t1/2 | Pre-dose(0h), 1, 2, 3, 4, 5, 6, (7), 8, 10, 12, 24, 48, 72, 96, 120 h
  16 times(fasting), 15 times(fed)

CONTACTS AND LOCATIONS:
Overall Officials: Kyungsoo Park, Ph D, MD, Principal Investigator — Yonsei University

REFERENCES:
- [Derived] Chae DW, Son H, Guk J, Park C, Park K. Pharmacokinetics of a nanocrystal-containing megestrol acetate formulation: a single-dose, randomized, open-label, 2-part, 2-period crossover study in healthy Korean subjects. Int J Clin Pharmacol Ther. 2016 Sep;54(9):698-704. doi: 10.5414/CP202574. PMID 27191767